CLINICAL TRIAL: NCT07290166
Title: A Phase II Study to Evaluate the Efficacy and Safety of Anti-HER2 Triple-targeted Drugs Combined With CDK4/6 Inhibitors in Neoadjuvant Therapy for ER-positive HER2-positive Breast Cancer Patients.
Acronym: Cinderella-Neo
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCHBCC-N098
Record Dates: First submitted 2025-12-06; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: ER positive and HER2 positive; triple-targeted anti-HER2 strategy; chemotherapy-free; neoadjuvant
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- triple-targeted anti-HER2 (Experimental): trastuzumab, pertuzumab, and pyrotinib combined with CDK4/6 inhibitor and endocrine therapy
  Interventions: Drug: triple-targeted anti-HER2 and CDK4/6 inhibitor

INTERVENTIONS:
Drug: triple-targeted anti-HER2 and CDK4/6 inhibitor — trastuzumab, pertuzumab, and pyrotinib combined with CDK4/6 inhibitor and endocrine therapy

SUMMARY:
To further enhance treatment efficacy, minimize reliance on chemotherapy, and identify the optimal neoadjuvant approach for ER-positive and HER2-positive population, we have designed a single-arm, phase II clinical trial. This study aims to evaluate the efficacy and safety of a novel regimen integrating CDK4/6 inhibitors intensified endocrine therapy and dual HER2-targeted monoclonal antibodies plus the tyrosine kinase inhibitor pyrotinib.

DETAILED DESCRIPTION:
In patients with ER-positive and HER2-positive breast cancer, the therapeutic potential of combining trastuzumab, pertuzumab, and pyrotinib-representing a triple-targeted anti-HER2 strategy-alongside intensified endocrine therapy( with CDK4/6 inhibitors )has not yet been established. To further enhance treatment efficacy, minimize reliance on chemotherapy, and identify the optimal neoadjuvant approach for this patient population, we have designed a single-arm, phase II clinical trial. This study aims to evaluate the efficacy and safety of a novel regimen integrating CDK4/6 inhibitors intensified endocrine therapy and dual HER2-targeted monoclonal antibodies plus the tyrosine kinase inhibitor pyrotinib.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18 to 70 years with breast cancer eligible for neoadjuvant therapy
2. Clinically staged as II-III
3. Histologically confirmed unilateral invasive breast cancer with HER2 positivity, defined as HER2 immunohistochemistry 3+ or in situ hybridization (FISH)-confirmed amplification
4. Estrogen receptor (ER) expression ≥10% by immunohistochemistry
5. Postmenopausal status
6. Premenopausal or perimenopausal patients must undergo surgical oophorectomy or receive ovarian function suppression with gonadotropin-releasing hormone (GnRH) agonists
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
8. Left ventricular ejection fraction (LVEF) ≥50% and corrected QT interval (QTc) ≤470 ms
9. Adequate major organ function, as evidenced by the following laboratory parameters:

(1) Hematologic function: hemoglobin (Hb) ≥90 g/L (without transfusion within 14 days), absolute neutrophil count (ANC) ≥1.5×10⁹/L, platelet count (PLT) ≥100×10⁹/L; (2) Hepatic and renal function: total bilirubin (TBIL) ≤1.5×upper limit of normal (ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3×ULN, serum creatinine ≤1×ULN, and calculated creatinine clearance >50 mL/min using the Cockcroft-Gault formula 10) Willingness to participate in the study, provision of signed informed consent, and demonstrated ability to comply with study procedures and follow-up visits

Exclusion Criteria:

1. HER2-negative disease, defined as immunohistochemistry (IHC) score of 0 or 1+; or IHC 2+ without amplification by fluorescence in situ hybridization (FISH)
2. Prior receipt of neoadjuvant therapy or any systemic or non-surgical local treatment, including chemotherapy, targeted therapy, radiotherapy, or endocrine therapy
3. History of another malignancy, except for adequately treated basal cell carcinoma of the skin or cervical carcinoma in situ
4. Inflammatory breast cancer, bilateral breast cancer, or presence of distant metastases
5. Pregnant or breastfeeding women, or women of childbearing potential who are unwilling or unable to use effective contraception during the study period
6. Concurrent participation in another interventional clinical trial
7. Significant organ dysfunction, including cardiac, pulmonary, hepatic, or renal impairment; left ventricular ejection fraction (LVEF) <50% on echocardiography; history of major cardiovascular or cerebrovascular events within 6 months prior to enrollment (e.g., unstable angina, chronic heart failure, myocardial infarction, or stroke); uncontrolled hypertension (>150/90 mmHg); or poorly controlled diabetes mellitus
8. Current use of strong CYP3A4 inhibitors or inducers, including:

   1. Strong inhibitors: boceprevir, clarithromycin, conivaptan, delavirdine, indinavir, itraconazole, ketoconazole, ritonavir, mibefradil, miconazole, trazodone, nelfinavir, posaconazole, saquinavir, telaprevir, telithromycin, voriconazole, grapefruit, grapefruit juice, or grapefruit-containing products
   2. Strong inducers: carbamazepine, phenytoin, primidone, rifampicin, and St. John's wort
9. Active, severe, or uncontrolled infection, or fever of unknown origin during the screening period
10. History of substance abuse involving psychotropic agents with ongoing dependence, or history of significant psychiatric disorder that may impair compliance or safety
11. Deemed unsuitable for study participation by the treating investigator

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
pCR | 3 years
  pathological response rate

SECONDARY OUTCOMES:
EFS | 3 years
  Event free survival
iDFS | 3 years
  invasive disease free survival
RFS | 3 years
  Recurrence free survival
DDFS | 3 years
  distant disease free survival
OS | 3 years
  overall survival
adverse events | 3 years
  adverse events according to CTCAE 5.0

IPD SHARING:
Plan to Share IPD: No